CLINICAL TRIAL: NCT05799391
Title: Efficacy of Soothing Cream Jel in Improving the Range of Motion and Chronic Pain at Shoulder and Elbow: A Double-blinded, Randomized, Placebo-Controlled Trial
Brief Title: RCT for the Efficacy of Soothing Cream Jel in Improving Upper Limb Pain and Motion
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCJ study
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Upper Extremity Problem

STUDY DESIGN:
Intervention Model Description: Soothing cream jel or placebo cream jel
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Soothing cream jel) (Experimental): Soothing cream jel
  Interventions: Drug: SJC
- Placebo (Placebo Comparator): Placebo cream jel
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SJC — Soothing cream jel
  Other Names: Soothing cream jel
  Arms: Active treatment (Soothing cream jel)
Other: Placebo — Placebo cream jel
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled clinical trial. This trial is used to evaluate the efficacy of soothing cream jel on chronic upper limb pain and the range of motion.

DETAILED DESCRIPTION:
Potential subjects will be screened according to the eligibility criteria after signing the informed consent form. Subjects who fulfill the requirements will be randomized into either the treatment group or the placebo group. And receive either soothing cream jel or placebo cream jel for 2 weeks. Then followed by a post-treatment for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60;
2. Participates in regular physical activity, at least once a week for 30 minutes;
3. Chronic pain in the shoulder or elbow longer than 3 months;
4. 11-items Numeric pain rating scale ≥4; and
5. Willing to provide written informed consent.

Exclusion Criteria:

1. The patient had received previous physiotherapy, acupuncture, Tui Na massage, or bone-setting treatment for distal upper limb pain within the past 2 weeks;
2. The pain was due to a fracture or known complex regional pain syndrome.
3. History of upper limb surgery;
4. Known severe medical conditions (e.g. rheumatoid arthritis, osteoporosis, cardiac, renal, hepatic, hematological diseases, vertigo, seizure, infection, malignancy, neurological impairment);
5. Concomitant drugs of NSAIDs, any kind of painkillers, or anti-inflammatory drugs 15 days prior to randomization;
6. Known impaired hematological profile and liver / renal function;
7. Known allergic history to any topical cream;
8. Known pregnant or lactating; or
9. Unable to complete questionnaires

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change of the range of motion | From baseline to week 2
  The range of motion of upper (shoulder or elbow) will be measured by a digital goniometer.
  For the shoulder, active flexion and abduction ROMs are measured using a goniometer while the participants are standing. For the elbow, both flexion and extension will be measured by a goniometer in a standing position.

SECONDARY OUTCOMES:
Chang of the range of motion | From baseline to week 4
  The range of motion of upper (shoulder or elbow) will be measured by a digital goniometer.
  For the shoulder, active flexion and abduction ROMs are measured using a goniometer while the participants are standing. For the elbow, both flexion and extension will be measured by a goniometer in a standing position.
Change of Numeric pain rating scale (NPRS) | 2 weeks
  It contains 11 items in which subjects select a whole number (0-10 integers) that best reflects the average intensity of subjects' pain in the past week. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Change of Numeric pain rating scale (NPRS) | 4 weeks
  It contains 11 items in which subjects select a whole number (0-10 integers) that best reflects the average intensity of subjects' pain in the past week. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Handgrip strength | 2 weeks
  Handgrip strengths are measured by a dynamometer, on the dominant hand of the participant. Participants are instructed to hold the device with the arm at the right angle and elbow to the side of the body. The maximum effort will be taken from three attempts.
Handgrip strength | 4 weeks
  Handgrip strengths are measured by a dynamometer, on the dominant hand of the participant. Participants are instructed to hold the device with the arm at the right angle and elbow to the side of the body. The maximum effort will be taken from three attempts.
Back-scratch test | 2 weeks
  The back-scratch test is used to measure the overall shoulder ROM. It is performed by measuring the distance between (or the overlap of) the middle fingers of both hands behind the back with a ruler.
Back-scratch test | 4 weeks
  The back-scratch test is used to measure the overall shoulder ROM. It is performed by measuring the distance between (or the overlap of) the middle fingers of both hands behind the back with a ruler.
Score change of American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASESp-S) | 2 weeks
  The ASESp-S consists of 18 questions from 3 sections: pain, instability and activities of daily living (ADL). Among the 18 questions, 11 self-report items represented functional ADL dimension (10 items) and pain dimension (1 item). The ADL section was scored on a 4-points-graded ordinal scale, ranging from 0 (unable to do) to 3 (not difficult) and cumulative scores were collected. The pain section was derived from the 10-points-graded visual analog scale (VAS) ranging from 0 (no pain) to 10 (maximum pain).
Score change of American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASESp-S) | 4 weeks
  The ASESp-S consists of 18 questions from 3 sections: pain, instability and activities of daily living (ADL). Among the 18 questions, 11 self-report items represented functional ADL dimension (10 items) and pain dimension (1 item). The ADL section was scored on a 4-points-graded ordinal scale, ranging from 0 (unable to do) to 3 (not difficult) and cumulative scores were collected. The pain section was derived from the 10-points-graded visual analog scale (VAS) ranging from 0 (no pain) to 10 (maximum pain).
Score change of American Shoulder and Elbow Surgeons Standardized Elbow Assessment Form (ASESp-E) | 2 weeks
  The ASESp-E consists of 3 sections: pain, function, and satisfaction. Patients are asked about the spot of pain in their elbow and asked to rate pain on a visual analog scale (VAS) in different situations, such as the worst of pain, at rest, lifting a heavy object, doing a task with repeated elbow movements and at night. The VAS ranges from 0 (no pain) to 10 (maximum pain). In the function section, patients are asked to rate their ability to perform 10 ADL and their usual work and sporting activities with the scale from 0 (unable to do) to 3 (not difficult).
Score change of American Shoulder and Elbow Surgeons Standardized Elbow Assessment Form (ASESp-E) | 4 weeks
  The ASESp-E consists of 3 sections: pain, function, and satisfaction. Patients are asked about the spot of pain in their elbow and asked to rate pain on a visual analog scale (VAS) in different situations, such as the worst of pain, at rest, lifting a heavy object, doing a task with repeated elbow movements and at night. The VAS ranges from 0 (no pain) to 10 (maximum pain). In the function section, patients are asked to rate their ability to perform 10 ADL and their usual work and sporting activities with the scale from 0 (unable to do) to 3 (not difficult).
Score change of 36-Item Short Form Survey (SF-36v2) | 2 weeks
  SF36 is a generic instrument to measure general health status. It will be used to assess the patient's health status using 8 different dimensions including vitality, physical functioning, bodily pain, general health perceptions, role limitations due to physical health, role limitations due to emotional health, social role functioning and mental health. The possible score ranges from 0 to 100 points whereby 0 points represent the greatest possible limitation of health, while 100 points represent the absence of health restrictions.
Score change of 36-Item Short Form Survey (SF-36v2) | 4 weeks
  SF36 is a generic instrument to measure general health status. It will be used to assess the patient's health status using 8 different dimensions including vitality, physical functioning, bodily pain, general health perceptions, role limitations due to physical health, role limitations due to emotional health, social role functioning and mental health. The possible score ranges from 0 to 100 points whereby 0 points represent the greatest possible limitation of health, while 100 points represent the absence of health restrictions.
Rescue drugs or treatments used for pain symptoms | From baseline to week 4
  If participants used any other drugs or treatments for the pain symptom during the whole study period, those drug names or treatments would be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, Principal Investigator — Hong Kong Institute of Integrative Medicine
Locations (1):
- Hong Kong Institute of Integrative Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and the statistical analysis plan are available after completion of the study and reporting of the results.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the study and reporting of the results.
Access Criteria: The principal investigator of this trial will be responsible for accessing the request.

REFERENCES:
- [Derived] Lo CW, Sum KWR, Leung FLE, Yang Y, Chan KL, Lam KK, Lau KW, Sum CH, Lin WL, Ho SH, Lin ZX. Efficacy of soothing cream gel in the range of motion and chronic pain at the shoulder and elbow: protocol of a double-blinded, randomised, placebo-controlled trial. BMJ Open. 2024 Jul 5;14(7):e085856. doi: 10.1136/bmjopen-2024-085856. PMID 38969378